CLINICAL TRIAL: NCT00520559
Title: Incidence of Cardiac Complications in Patients With Cardiac Siderosis During 1 Year Follow-up and the Normal T2* Ranges in LVF, MI and Normal Population.
Brief Title: T2* in Transfusion Dependant Anemia, MI, LVF, Normal Patients
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Other Study IDs: 07/MRE04/32
Record Dates: First submitted 2007-08-23; First posted 2007-08-24 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Thalassemia
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thalassemia

SUMMARY:
The purpose of this study is to provide accurate prognostic data linking cardiac complications to myocardial T2* values (A measure of iron levels in the heart using MRI)in patients predisposed to heart iron overload.

DETAILED DESCRIPTION:
Key Definitions Myocardial siderosis - Iron deposition that occurs in the heart, usually in relation to recurrent blood transfusions and red cell breakdown.

Thalassaemia - A hereditary form of anaemia leading to recurrent blood transfusions and iron overload.

Cardiomyopathy - Disease of the heart leading to heart failure. In the case of cardiac siderosis it is entirely reversible.

Chelation - Drug used to remove iron from the heart T2* CMR - Cardiac Magnetic Resonance Imaging. A specialised scan that uses a large magnet to image the heart. As iron has magnetic properties we can use this scan to determine the amount of iron within the heart. T2* is a value that relates to the level of iron loading in the heart. A T2* of less than 10 relates to severe heart iron loading, a T2* of 10-20 relates to mild/moderate heart iron loading and a T2* of greater than 20 relates to no significant iron loading in the heart.

Heart failure - Disease in which the myocardium (heart muscle) weakens and can not pump blood efficiently. Fluid accumulates in the lungs, hands, ankles, or other parts of the body. The mortality from heart failure is very high.

Heterozygotes - An individual with one normal and one abnormal thalassaemia gene. They are carriers of the thalassaemia gene with milder clinical manifestations.

Homozygotes - An individual who has inherited both abnormal thalassaemia genes producing a more severe form of the disease.

Question Response Although a rare disease in the UK, thalassaemia is the commonest genetic disorder worldwide, with approximately 94 million heterozygotes for beta thalassaemia and 60,000 homozygotes born each year.

In the United Kingdom, despite relatively easy access to healthcare, approximately 50% of patients with thalassaemia major die before reaching the age of thirty five. Of those deaths, over 60% are a result of heart failure. The cardiomyopathy is reversible if chelation is commenced early but diagnosis is often delayed due to the late onset of symptoms and measurable LV dysfunction.

This study will provide strong evidence that a myocardial T2* <10ms represents a high risk of developing cardiac complications. Derived risk ratios will provide sound guidance as to when life saving chelation is required.

A database will be produced containing clinical data and T2* values on 665 thalassaemia patients from 1998-2006.

A diagnosis of heart failure will be made if the patient has had an ejection fraction of less than 55% (measured by CMR or echocardiography) and symptoms as per NHYA classification within 1 year of their CMR scan.

A diagnosis of arrhythmia was made if the patient had documented ECG evidence within 1 year of their CMR scan.

This information will be gathered retrospectively by access to outpatient clinic letters, hospital notes, CMR/ echo reports and clinical details recorded in a proforma at the time of the CMR scan. Some of the clinical data would be obtained from other hospitals.

Patient scans will only be used if between the dates of 1999-2005. As all other data is in respect to the year immediately post scan then no further data will be required on any patient post 2006.

Logistic regression will be used to determine whether T2* is predictive of cardiac complications in the 12 months after a patient's CMR scan. Since some patients will have more than 1 scan, a mixed model logistic regression will be used to take account of any within-patient correlation that may occur.

The data will be analysed by Dr Michael Roughton (Medical Statistician, Royal Brompton Hospital)

The results will be disseminated through peer review journals

ELIGIBILITY:
Inclusion Criteria:

* Thalassaemia Major
* Patient must have had a cardiac MRI scan between 1999 and 2006

Exclusion Criteria:

* Other structural heart disease such as valvular abnormalities, MI, congenital heart disease

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Please note that the age range detailed above refers to the normal group (63 patients): the study article provided by the study team to complete this record only provides a mean age range for the 39 Left Ventricular Dysfunction Group (50.1 +/- 14.0 years) and 24 Septal Infarction Group (58.6 +/- 13.9).
Sampling Method: Non-Probability Sample
Enrollment: 652 (Actual)
Dates: Start 2007-01; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Heart Failure | 1yr
  Ejection fraction
Arrhythmia | 1yr
  ECG

CONTACTS AND LOCATIONS:
Overall Officials: Dudley Pennell, MA, MD, Principal Investigator — Imperial College London

REFERENCES:
- [Result] Kirk P, Roughton M, Porter JB, Walker JM, Tanner MA, Patel J, Wu D, Taylor J, Westwood MA, Anderson LJ, Pennell DJ. Cardiac T2* magnetic resonance for prediction of cardiac complications in thalassemia major. Circulation. 2009 Nov 17;120(20):1961-8. doi: 10.1161/CIRCULATIONAHA.109.874487. Epub 2009 Oct 2. PMID 19801505
- [Derived] Kirk P, Sheppard M, Carpenter JP, Anderson L, He T, St Pierre T, Galanello R, Catani G, Wood J, Fucharoen S, Porter JB, Walker JM, Forni GL, Pennell DJ. Post-mortem study of the association between cardiac iron and fibrosis in transfusion dependent anaemia. J Cardiovasc Magn Reson. 2017 Mar 27;19(1):36. doi: 10.1186/s12968-017-0349-3. PMID 28343449
- [Derived] Kirk P, He T, Anderson LJ, Roughton M, Tanner MA, Lam WW, Au WY, Chu WC, Chan G, Galanello R, Matta G, Fogel M, Cohen AR, Tan RS, Chen K, Ng I, Lai A, Fucharoen S, Laothamata J, Chuncharunee S, Jongjirasiri S, Firmin DN, Smith GC, Pennell DJ. International reproducibility of single breathhold T2* MR for cardiac and liver iron assessment among five thalassemia centers. J Magn Reson Imaging. 2010 Aug;32(2):315-9. doi: 10.1002/jmri.22245. PMID 20677256